CLINICAL TRIAL: NCT06083740
Title: A Postmarket Clinical Follow Up Study (PMCF) to Evaluate the Safety and Performance of VERIFORTE/Granudacyn® Med Wound Irrigation Solution.
Status: Completed | Type: Observational
Sponsor: P.G.F. Industry Solutions GmbH (Industry)
Collaborators: WPM - Wund Pflege Management Ges.m.b.H (Unknown)
Responsible Party: Sponsor
Other Study IDs: CIP_WSL_2022_001
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Wounds
Keywords: Acute wounds, chronic wounds, burns
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Granudacyn/Veriforte — Wound irrigation solution for all kinds of wounds (Acute, chronic or contaminated wounds).

SUMMARY:
In the course of this clinical trial, it was shown that the use of Granudacyn/VERIFORTE med wound irrigation solution in the course of adjuvant therapy supports wound healing through mechanical irrigation and moistening of the wound. No risks have been reported. The benefits of using Granudacyn/VERIFORTE med wound irrigation solution therefore outweigh the potential risks.

DETAILED DESCRIPTION:
Aim of this clinical trial was to collect clinical data on the performance and safety of the use of Granudacyn/VERIFORTE med as a wound irrigation solution, for cleansing and irrigation of acute, chronic or contaminated wounds.

The evaluation of the safety of the use of Granudacyn/VERIFORTE med wound irrigation solution within the scope of use was based on the frequency of adverse events (AEs) and, in particular, treatment-emergent adverse events (ADEs).

Study Design:

* Open-label, retrospective, monocentric, PMCF, non-interventional, observational study.
* One treatment group (single arm): All subjects participating in the study will be treated with Granudacyn/VERIFORTE med wound irrigation solution.
* The study will be conducted in Austria. The participating trial centre is in Lower Austria: WPM Ges.m.b.H

ELIGIBILITY:
Inclusion Criteria:

* Presence of a documented case report within the indication, which enables a retrospective evaluation of the target variables.
* Subjects are ≥ 18 years of age.
* Gender: All.

Exclusion Criteria:

* Vulnerable persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One treatment group (single-arm): All subjects participating in the study will be treated with Granudacyn/VERIFORTE med wound irrigation solution. People with a completed treatment of an acute or chronic wound participated in the study.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety: • AES: 0,00%, 95% CI: (0,00% - 4,16%) • ADEs: 0,00%, 95% CI: (0,00% - 4,16%) | 9 months
  Evaluation of the safety of the use of Granudacyn/VERIFORTE med wound irrigation solution within the scope of use, based on the frequency of adverse events (AEs) and, in particular, treatment-emergent adverse events (ADEs).

CONTACTS AND LOCATIONS:
Locations (1):
- PGF Industry Solutions GmbH, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No